CLINICAL TRIAL: NCT02560064
Title: Length of Small Bowel. How Can Standardise Measurement and Why?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Servet Karagül, medical doctor, Inonu University
Other Study IDs: 2015/114
Record Dates: First submitted 2015-09-16; First posted 2015-09-25 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Small/Large Bowel
MeSH Terms: conditions — Cerebral Palsy | interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- laparotomy and small bowel length: measurement of small bowel length in laparotomies
  Interventions: Procedure: Laparotomy

INTERVENTIONS:
Procedure: Laparotomy — Small bowel length will measure in laparotomy, regardless of indication.

SUMMARY:
Measurement of the small bowel length studied by anatomists, surgeons and radiologists. Results were highly different among these series. Technical and mechanical factors have major effects on measures. Investigators decided to reach a standardization for the measurement of small bowel length.

DETAILED DESCRIPTION:
Small bowel length will be measure in patients undergoing intraabdominal surgery. This will be establish by two surgeon from Treitz ligament to ileocecal valve two, consecutively. For measurement, a tape will place to antimesenteric, mesenteric border and the midline between these two sides.

Exclusion criteria include patients with inflammatory bowel disease, peritonitis, prior abdominal surgery.

Demographic data, patients clinical details and small bowel length will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for abdominal surgery

Exclusion Criteria:

* Inflammatory bowel disease
* History of intraabdominal surgery
* peritonitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Power analyse was done. Study include at least 44 patients.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Length of Small Bowel. How Can Standardise Measurement and Why? | postop 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt Kayaalp, Study Director — Inonu University, Faculty of Medicine